CLINICAL TRIAL: NCT03037177
Title: Mediastinal Grey Zone Lymphoma: Clinico-pathological Characteristics and Outcomes of 99 Patients From the LYSA
Brief Title: Mediastinal Grey Zone Lymphoma From the LYSA
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0721
Record Dates: First submitted 2016-11-04; First posted 2017-01-31 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2016-10

CONDITIONS: Mediastinal Grey Zone Lymphoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — clinical characteristics and outcomes of a large retrospective series of 99 cases centrally reviewed by a panel of hematopathologists.

GROUPS / COHORTS (3):
- CHL like GZL: Classical Hodgkin Lymphoma like Grey Zone Lymphoma (morphology of CHL and phenotype of PMBCL)
- PMBCL like GZL: Primary Mediastinal B Cell Lymphoma like Grey Zone Lymphoma(morphology of PMBCL and phenotype of CHL)
- Composite: with a morphology of CHL on the one side and of PMBCL on the other side of the same diagnosis biopsy

SUMMARY:
Mediastinal grey zone lymphoma, B cell lymphomas with intermediate features between classical Hodgkin lymphoma and primary mediastinal B cell lymphoma, are not well described in the literature. Investigators report the clinical characteristics and outcomes of a large retrospective series of 99 cases centrally reviewed by a panel of hematopathologists, with a consensus established for the diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* cases with an intermediate morphology and phenotype between CHL and PMBCL were included after central pathological review

Exclusion Criteria:

* Cases of CHL with partial CD20 expression or low expression in tumoral cells were excluded and considered as CD20-positive CHL
* Exclusion of sequential form patients (with a diagnostic biopsy of PMBCL and a relapse biopsy of CHL or vise-versa) as they represent a biases for statistical analysis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We retrospectively identified cases treated in French, Belgium and Portuguese LYSA centers suspected to be MGZL using local pathological records, records from LYSA centers and the LYMPHOPATH network, which aims to review all newly diagnosed lymphoma cases in France (14). All the FFPE blocks and immunohistochemistry (IHC) slides (obtained prior any treatment) were centralized in the LYSA-Pathology (LYSA-P) department located in Henri Mondor hospital in Paris to perform a central review by a panel of hematopathologists. Two hundred and four cases were reviewed by the panel of LYSA hematopathologists.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2013-01; Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
EFS in the global population of GZL | EFS: Event Free Survival from date of randomization until the date of first documented progression, up to 130 months
  Event-free survival (EFS) was calculated from the date of diagnosis to the date of progression, a change of therapy that was not initially scheduled (radiotherapy, high-dose therapy with autologous stem cell transplantation and other unplanned treatments) or death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre hospitalier Lyon sud, Pierre-Bénite, Auvergne-Rhône-Alpes, France